CLINICAL TRIAL: NCT05465655
Title: Pilot Study to Estimate a Reduction of TAVR Associated Conduction Disturbance Through Notification of Cara Monitor During TAVR Procedure
Brief Title: Cara CDRM (Conduction Disturbance Risk Monitor) 2.0
Acronym: Cara CDRM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment rate
Sponsor: Cara Medical Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Cara 2.0
Record Dates: First submitted 2022-07-15; First posted 2022-07-20 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2023-08

CONDITIONS: Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients undergoing TAVR (Experimental): Study subjects will be studied during the TAVR procedure and their 12 lead ECGs collected and analyzed notifying for New-Onset Conduction Disturbances (NOCD) using Cara Monitor.
  Interventions: Other: ECG monitoring for Conduction Disturbances

INTERVENTIONS:
Other: ECG monitoring for Conduction Disturbances — Continuous ECG monitoring of Conduction Disturbances in patients undergoing TAVR procedure
  Other Names: Continues ECG monitoring

SUMMARY:
Prospective, multicenter, roll-in, pilot clinical trial.

Study subjects will be studied during the TAVR procedure and their 12 lead ECGs collected and analyzed for New-Onset Conduction Disturbances (NOCD).

The study will be conducted in two stages:

During the first roll-in stage of the study, 50 intended to undergo TAVR (all comers) will be enrolled.

Data will be collected according to the study schedule below of pre-, during and after the TAVR procedure up to 14 days FU.

This data for the first 50 patients will be analyzed to evaluate the ability of the Cara Monitor prediction of NOCD post TAVR.

The second stage of the stage will be conducted upon completion of the first stage analysis and will be considered to randomize 1:1 the subjects connected to Cara Monitor during the procedure versus site-specific current practice.

The effect of Cara Monitor on reduction of NOCD post TAVR compared to patients treated and followed per regular site-specific practice will be estimated.

DETAILED DESCRIPTION:
Data to be collected during the study procedure for both stages:

1. Pre-procedure:

   1. Demographics, medical history, cardiac history, medications
   2. Cardiac CT raw data to be collected from all the pre-procedure CT scans performed in Medical Centers and from out-of-hospital sources (if available).
   3. In hospital 12 lead ECG
2. Procedure:

   During the procedure, the 12 lead ECG will be recorded processed, and displayed on the Cara monitor that is connected to Norav NR-1207-3 ECG Holter System. The Hemodynamic and Fluoroscopy monitors will be recorded on a commercially available video recorder.
3. Post-procedure (in hospital)

   1. After the procedure patients will continue to be connected to a commercially available to a commercially available 14 days ambulatory Holter monitor (AEM) (e.g. Bittium Faros™ ; MoMe™ Kardia) and will remain with the patient after the discharge for 14 days.
   2. Hospital standard 12 lead ECG will be recorded after the procedure, downloaded and collected by the study team.
4. Post-procedure - out of hospital:

   At discharge, patients will stay connected to the ambulatory Holter monitor (AEM) (Bittium Faros™; MoMe™ Kardia ) for 14 days post-procedure. Holter will be collected from patients at the end of the 14-day recording and its data downloaded and collected.

   Patients will be followed according to the current medical practice.
5. Follow-up according to the current medical practice a. 30 days follow-up hospital visit: i. Cardiac echo (if available) ii. 12 lead ECG b. 6 month - Clinical FU phone call c. 12 months Clinical FU phone call

Conduction Disturbances (CD) outcome will be subdivided into:

1. PPM or High-Grade AV Block (HGAVB)
2. All other new onset (or deterioration) of CD that are not listed in #1
3. No new onset CD

ELIGIBILITY:
Inclusion Criteria:

1. Must meet be ≥ 18 years of age.
2. Must meet indications for TAVR using approved devices
3. Provided written informed consent as approved by the Institutional Review Board (IRB) of the respective clinical site.
4. Willing to comply with specified follow-up evaluations.
5. Must meet the legal minimum age to provide Informed Consent based on local regulatory requirements.

Exclusion Criteria:

1. Any implanted device or an indication for treatment with rhythm management device (i.e., pacemaker, Cardiac Resynchronization Therapy (CRT) or Cardiac Resynchronization Therapy with cardioverter-defibrillator (CRT-D) at baseline.
2. Any contraindication to the TAVR procedure according to the instructions for use.
3. Less than the legal age of consent, legally incompetent, or otherwise vulnerable.
4. Planned treatment with any other investigational device, drug, or procedure (excluding registries) during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Evaluate Cara performance in reduction of New Onset Conduction Disturbances (NOCD) | 14 days
  Estimate the reduction of NOCD (percentage) at 14 days post TAVR while using Cara Monitor
Evaluate Cara performance in reduction of Permanent Pacemaker (PPM) or High-Grade AV Block (HGAVB) | 14 days
  Estimate the reduction (a percentage) of PPM or High-Grade AV Block (HGAVB)
Evaluate Cara usability using a dedicated questioner | 1 Day of Procedure
  Estimate learning curve of using CaraTM system (e.g. the experience required with system for achieving above improvements)
Evaluate Cara Safety, collecting Adverse Events | 14 days
  During the study patients will be followed for any adverse events relevant to the TAVR procedure as defined in the CRF

CONTACTS AND LOCATIONS:
Overall Officials: Helena Grinberg, PhD, Study Chair — Cara Medical Ltd
Locations (1):
- Mackram F. Eleid, M.D., Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No